CLINICAL TRIAL: NCT00748566
Title: A One-Year, Phase IV, Open-Label, Non-Comparative Trial Of The Effect Of Ziprasidone HCL On Metabolic Syndrome Risk Factors In Patients With Psychotic Disorders
Brief Title: One-Year Trial Of Oral Ziprasidone In Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281173
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia and Disorders With Psychotic Features
Keywords: Ziprasidone; metabolic syndrome; risk factors; schizophrenia; psychotic disorders.
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Metabolic Syndrome; Schizophrenia; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (switch to oral Ziprasidone) (Experimental)
  Interventions: Drug: Ziprasidone HCL (oral)

INTERVENTIONS:
Drug: Ziprasidone HCL (oral) — Ziprasidone Hydrochloride 20 to 80 mg administered orally twice a day (40 to 160 mg total daily dose) for up to 1 year.
  Other Names: Zeldox, Geodon

SUMMARY:
The purpose of this study is to explore the impact of ziprasidone on the distribution of metabolic syndrome risk factors in a population of patients presenting with glucose intolerance, dyslipidemia and/or elevated waist circumference associated with their current antipsychotic medication.

DETAILED DESCRIPTION:
The trial was terminated prematurely on May 24, 2012, due to changes in organizational strategy and resources. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subject must present at least 2 of the following risk factors of MS at screening: Elevated waist circumference: >102 cm in men and >88 cm in women; Elevated triglycerides (TGs): ≥1.7 mmol/L (≥150 mg/dL); Reduced HDL-Cholesterol: <1.03 mmol/L (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women; Elevated fasting glucose: ≥ 5.6 mmol/L.
* According to the clinical judgment of the investigator, the risk factors for MS have developed in close temporal relationship to starting an antipsychotic medication.
* Substitution to a less metabolically disruptive antipsychotic medication is considered.

Exclusion Criteria:

* Subjects with contraindication(s) to the use of Ziprasidone according to Canadian prescribing information.
* Subjects with a history of treatment resistance.
* Subjects with any medical condition (e.g. pre-existing diabetes, pre-existing dyslipidemia, thyroid pathology) or taking any concomitant medication (e.g. topiramate or other weight loss-promoting agents, hypoglycemic agents, hypolipemic agents), that may confound the evaluation of the study drug.
* Body mass index ≥ 40 at baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- Canada (23):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Medicine Hat, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Penticton, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Chatham, Ontario
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Markham, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Verdun, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Chue P, Mandel FS, Therrien F. The effect of ziprasidone on metabolic syndrome risk factors in subjects with schizophrenia: a 1 year, open-label, prospective study. Curr Med Res Opin. 2014 Jun;30(6):997-1005. doi: 10.1185/03007995.2014.898139. Epub 2014 Mar 17. PMID 24568177
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281173&StudyName=One-Year%20Trial%20Of%20Oral%20Ziprasidone%20In%20Patients%20With%20Metabolic%20Syndrome

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone: Ziprasidone 40 milligram (mg) capsule orally twice daily from Day 1 to 3, followed by ziprasidone 60 mg capsule orally twice daily from Day 4 to 7, then ziprasidone 80 mg capsule orally twice daily from Day 8 to 15 and thereafter ziprasidone 20 to 80 mg capsule orally twice daily as per investigator's discretion from Day 16 to 365.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 172
Completed | 60
Not Completed | 112
Not completed — Adverse Event | 49
Not completed — Death | 1
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 13
Not completed — Withdrawal by Subject | 22
Not completed — Study terminated by sponsor | 5
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Groups:
- Ziprasidone: Ziprasidone 40 mg capsule orally twice daily from Day 1 to 3, followed by ziprasidone 60 mg capsule orally twice daily from Day 4 to 7, then ziprasidone 80 mg capsule orally twice daily from Day 8 to 15 and thereafter ziprasidone 20 to 80 mg capsule orally twice daily as per investigator's discretion from Day 16 to 365.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least 1 Risk Factor Reduction From Baseline for Metabolic Syndrome (MS)
Description: MS risks factors: elevated (el) waist, men:>=102 centimeters(cm), women:>=88 cm (Asian origin:>=90 cm in men, >=80 cm in women); el triglycerides: >=1.7 millimoles per liter (mmol/L) (>=150 milligram per deciliter [mg/dL]); reduced high-density lipoprotein cholesterol (HDL-C), men:<1.03 mmol/L (<40 mg/dL), women:<1.3 mmol/L (<50 mg/dL); el fasting glucose: >=5.6 mmol/L (>=100 mg/dL); el systolic/diastolic blood pressure (SBP/DBP): SBP>=130 millimeters of mercury (mmHg) and/or DBP>=85 mmHg. Responder=at least 1 less risk factor at endpoint (premature discontinuation or Week 52) than baseline.
Time Frame: Endpoint (premature discontinuation or Week 52)
Population: Per protocol (PP) population included all enrolled participants who received at least 1 dose of study medication, had baseline and at least 1 post-baseline MS measure, and remained in the study for at least 16 weeks. Missing values were imputed using last observation carried forward (LOCF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
percentage of participants | 58.77 [47.0 to 71.0]

2. Secondary Outcome: Mean Change From Baseline in the Number of Risk Factors of Metabolic Syndrome (MS) at Week 4, 12, 28 and 52
Description: MS risks factors: elevated waist circumference: greater than or equal to (>=)102 cm in men, >=88 cm in women (Asian origin: >=90 cm [men], >=80 cm [women]); elevated triglycerides: >=1.7 mmol/L (>=150 mg/dL); reduced high-density lipoprotein cholesterol (HDL-C): less than (<)1.03 mmol/L (<40 mg/dL) in men, <1.3 mmol/L (<50 mg/dL) in women; elevated fasting glucose: >=5.6 mmol/L (>=100 mg/dL); elevated SBP/DBP: SBP >=130 mmHg and/or DBP >=85 mmHg.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: PP population. Missing values at Week 52 were imputed using LOCF. n=participants evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: risk factors
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
risk factors
  Baseline (n=114) | 3.4 (1.0)
  Change at Week 4 (n=113) | -0.3 (1.0)
  Change at Week 12 (n=112) | -0.4 (1.1)
  Change at Week 28 (n=98) | -0.7 (1.3)
  Change at Week 52 (n=114) | -0.8 (1.2)

3. Secondary Outcome: Percentage of Participants With Metabolic Syndrome (MS)
Description: According to the National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATPIII), metabolic syndrome is defined as a condition that includes 3 or more of 5 characteristics: abdominal obesity, hypertriglyceridemia, low high-density lipoprotein (HDL) cholesterol, high blood pressure, and high fasting glucose.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
percentage of participants
  Baseline (n=114) | 79.82 [71.6 to 88.1]
  Week 4 (n=113) | 70.80 [60.8 to 80.8]
  Week 12 (n=112) | 72.32 [62.6 to 82.1]
  Week 28 (n=98) | 58.16 [45.4 to 71.0]
  Week 52 (n=114) | 52.63 [40.0 to 65.3]

4. Secondary Outcome: Number of Participants With Change From Baseline in Metabolic Syndrome (MS) Risk Factors at Week 4, 12, 28 and 52
Description: MS risks factors: elevated waist circumference: >=102 cm in men, >=88 cm in women (Asian origin: >=90 cm [men], >=80 cm [women]); elevated triglycerides: >=1.7 mmol/L (>=150 mg/dL); reduced high-density lipoprotein cholesterol (HDL-C): <1.03 mmol/L (<40 mg/dL) in men, <1.3 mmol/L (<50 mg/dL) in women; elevated fasting glucose: >=5.6 mmol/L (>=100 mg/dL); elevated SBP/DBP: SBP >=130 mmHg and/or DBP >=85 mmHg.
Time Frame: Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
participants
  Week 4: Decrease by at least 1 risk factor (n=113) | 46
  Week 4: No change in risk factor (n=113) | 46
  Week 4: Increase by at least 1 risk factor (n=113) | 21
  Week 12:Decrease by at least 1 risk factor (n=112) | 44
  Week 12: No change in risk factor (n=112) | 51
  Week 12:Increase by at least 1 risk factor (n=112) | 17
  Week 28: Decrease by at least 1 risk factor (n=98) | 45
  Week 28: No change in risk factor (n=98) | 39
  Week 28: Increase by at least 1 risk factor (n=98) | 14
  Week 52:Decrease by at least 1 risk factor (n=114) | 67
  Week 52: No change in risk factor (n=114) | 35
  Week 52:Increase by at least 1 risk factor (n=114) | 12

5. Secondary Outcome: Percentage of Participants With Individual Risk Factors of Metabolic Syndrome (MS)
Description: as for outcome 4
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
percentage of participants
  Baseline: Elevated waist circumference (n=114) | 93.86 [89.3 to 98.4]
  Baseline: Elevated triglycerides (n=114) | 83.33 [75.8 to 90.8]
  Baseline: Reduced HDL-C (n=114) | 78.07 [69.5 to 86.7]
  Baseline: Elevated SBP (n=114) | 32.46 [17.4 to 47.5]
  Baseline: Elevated DBP (n=114) | 26.32 [10.6 to 42.1]
  Baseline: Elevated fasting glucose (n=114) | 44.74 [31.1 to 58.4]
  Week 4: Elevated waist circumference (n=113) | 88.50 [82.2 to 94.7]
  Week 4: Elevated triglycerides (n=111) | 60.36 [48.6 to 72.1]
  Week 4: Reduced HDL-C (n=113) | 71.68 [61.9 to 81.5]
  Week 4: Elevated SBP (n=113) | 31.86 [16.6 to 47.1]
  Week 4: Elevated DBP (n=113) | 29.20 [13.7 to 44.7]
  Week 4: Elevated fasting glucose (n=113) | 46.02 [32.5 to 59.6]
  Week 12: Elevated waist circumference (n=112) | 83.93 [76.5 to 91.4]
  Week 12: Elevated triglycerides (n=112) | 61.61 [50.1 to 73.1]
  Week 12: Reduced HDL-C (n=112) | 72.32 [62.6 to 82.1]
  Week 12: Elevated SBP (n=112) | 29.46 [13.9 to 45.0]
  Week 12: Elevated DBP (n=112) | 31.25 [15.9 to 46.6]
  Week 12: Elevated fasting glucose (n=112) | 36.61 [21.9 to 51.4]
  Week 28: Elevated waist circumference (n=100) | 76.00 [66.4 to 85.6]
  Week 28: Elevated triglycerides (n=99) | 56.57 [43.6 to 69.5]
  Week 28: Reduced HDL-C (n=99) | 61.62 [49.4 to 73.8]
  Week 28: Elevated SBP (n=100) | 29.00 [12.5 to 45.5]
  Week 28: Elevated DBP (n=100) | 35.00 [19.2 to 50.8]
  Week 28: Elevated fasting glucose (n=99) | 37.37 [21.8 to 53.0]
  Week 52: Elevated waist circumference (n=114) | 72.81 [63.2 to 82.4]
  Week 52: Elevated triglycerides (n=114) | 52.63 [40.0 to 65.3]
  Week 52: Reduced HDL-C (n=114) | 63.16 [52.0 to 74.3]
  Week 52: Elevated SBP (n=114) | 28.95 [13.5 to 44.4]
  Week 52: Elevated DBP (n=114) | 28.95 [13.5 to 44.4]
  Week 52: Elevated fasting glucose (n=114) | 32.46 [17.4 to 47.5]

6. Secondary Outcome: Change From Baseline in Waist Circumference at Week 4, 12, 28 and 52
Description: Waist circumference data is reported separately for male and female participants.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
cm
  Baseline: Male (n=79) | 110.8 (10.0)
  Baseline: Female (n=35) | 108.9 (10.5)
  Change at Week 4: Male (n=78) | -1.0 (3.1)
  Change at Week 4: Female (n=35) | 0.4 (3.0)
  Change at Week 12: Male (n=77) | -2.1 (4.9)
  Change at Week 12: Female (n=35) | -2.4 (6.8)
  Change at Week 28: Male (n=70) | -3.7 (7.2)
  Change at Week 28: Female (n=30) | -2.5 (5.8)
  Change at Week 52: Male (n=79) | -3.6 (7.5)
  Change at Week 52: Female (n=35) | -4.0 (8.9)

7. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at Week 4, 12, 28 and 52
Description: BP measurement is recorded as systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles).
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
mmHg
  Baseline: SBP (n=114) | 124.3 (13.3)
  Baseline: DBP (n=114) | 80.7 (9.5)
  Change at Week 4: SBP (n=113) | -1.0 (10.0)
  Change at Week 4: DBP (n=113) | -0.4 (7.6)
  Change at Week 12: SBP (n=112) | -1.0 (11.8)
  Change at Week 12: DBP (n=112) | -0.1 (8.0)
  Change at Week 28: SBP (n=100) | -1.0 (11.9)
  Change at Week 28: DBP (n=100) | 0.0 (9.5)
  Change at Week 52: SBP (n=114) | -1.0 (11.2)
  Change at Week 52: DBP (n=114) | -1.1 (8.8)

8. Secondary Outcome: Change From Baseline in Triglyceride and High Density Lipoprotein-Cholesterol (HDL-C) Levels at Week 4, 12, 28 and 52
Description: Triglyceride data is reported for whole study population whereas HDL-C data is reported separately for male and female participants.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
mg/dL
  Baseline: Triglyceride (n=114) | 242.8 (115.1)
  Baseline: HDL-C, Male (n=79) | 35.8 (7.2)
  Baseline: HDL-C, Female (n=35) | 41.9 (9.0)
  Change at Week 4: Triglyceride (n=111) | -37.3 (103.8)
  Change at Week 4: HDL-C, Male (n=78) | 1.2 (5.1)
  Change at Week 4: HDL-C, Female (n=35) | 2.1 (7.8)
  Change at Week 12: Triglyceride (n=112) | -39.5 (93.9)
  Change at Week 12: HDL-C, Male (n=77) | 2.1 (6.0)
  Change at Week 12: HDL-C, Female (n=35) | 1.8 (5.8)
  Change at Week 28: Triglyceride (n=99) | -52.3 (103.8)
  Change at Week 28: HDL-C, Male (n=69) | 3.1 (5.4)
  Change at Week 28: HDL-C, Female (n=30) | 4.5 (8.0)
  Change at Week 52: Triglyceride (n=114) | -60.0 (100.7)
  Change at Week 52: HDL-C, Male (n=79) | 3.9 (7.0)
  Change at Week 52: HDL-C, Female (n=35) | 5.0 (8.8)

9. Secondary Outcome: Change From Baseline in Fasting Glucose Level at Week 4, 12, 28 and 52
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
mg/dL
  Baseline (n=114) | 104.5 (25.7)
  Change at Week 4 (n=113) | -0.8 (19.7)
  Change at Week 12 (n=112) | -4.0 (20.3)
  Change at Week 28 (n=99) | -5.0 (19.1)
  Change at Week 52 (n=114) | -3.0 (31.0)

10. Secondary Outcome: Change From Baseline in 10-year Cardiovascular Heart Disease (CHD) Risk According to Framingham Scoring System at Week 4, 12, 28 and 52
Description: Framingham scoring system risk factors: age (risk points range: -9 to 16), cholesterol (risk points range: 0 to 13), HDL cholesterol (risk points range: -1 to 2), smoking (risk points range: 0 to 9), and systolic blood pressure (risk points range: 0 to 6); total risk points range <0 to >=25, higher score indicates higher CHD risk. The risk points are transformed to 10-year risk percentage for CHD which ranges from <1% to >=30%, where higher percent indicates greater risk for CHD.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: PP population. Missing values at Week 52 were imputed using LOCF. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: percent of 10-year CHD risk
Arm/Group | Ziprasidone
Number analyzed (Participants) | 113
percent of 10-year CHD risk
  Baseline (n=113) | 9.3 (5.9)
  Change at Week 4 (n=112) | -0.7 (2.5)
  Change at Week 12 (n=111) | -0.9 (2.1)
  Change at Week 28 (n=97) | -1.2 (2.3)
  Change at Week 52 (n=113) | -1.3 (2.4)

11. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) and Low Density Lipoprotein-Cholesterol (LDL-C) Levels at Week 4, 12, 28 and 52
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
mmol/L
  Baseline: TC (n=114) | 5.5 (1.1)
  Baseline: LDL-C (n=114) | 3.3 (1.1)
  Change at Week 4: TC (n=113) | -0.3 (0.8)
  Change at Week 4: LDL-C (n=110) | -0.1 (0.8)
  Change at Week 12: TC (n=112) | -0.4 (0.8)
  Change at Week 12: LDL-C (n=112) | -0.2 (0.8)
  Change at Week 28: TC (n=99) | -0.4 (0.8)
  Change at Week 28: LDL-C (n=97) | -0.2 (0.7)
  Change at Week 52: TC (n=114) | -0.5 (0.7)
  Change at Week 52: LDL-C (n=114) | -0.3 (0.8)

12. Secondary Outcome: Change From Baseline in Weight at Week 4,12, 28 and 52
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
kilogram (kg)
  Baseline (n=114) | 96.5 (16.9)
  Change at Week 4 (n=113) | -0.9 (3.9)
  Change at Week 12 (n=112) | -2.4 (5.1)
  Change at Week 28 (n=100) | -3.8 (7.4)
  Change at Week 52 (n=114) | -4.4 (8.4)

13. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 4, 12, 28 and 52
Description: Body mass index calculated as weight in kilograms (kg) divided by height in (meters) squared (m)^2 .
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
kg/m^2
  Baseline (n=114) | 32.4 (4.3)
  Change at Week 4 (n=113) | -0.3 (1.2)
  Change at Week 12 (n=112) | -0.8 (1.6)
  Change at Week 28 (n=100) | -1.2 (2.3)
  Change at Week 52 (n=114) | -1.5 (2.8)

14. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Concentration at Week 4, 12, 28 and 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, Week 4, 12, 28, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Ziprasidone
Number analyzed (Participants) | 114
percentage of total hemoglobin
  Baseline (n=114) | 5.7 (0.8)
  Change at Week 4 (n=111) | -0.0 (0.2)
  Change at Week 12 (n=112) | -0.0 (0.3)
  Change at Week 28 (n=99) | -0.1 (0.4)
  Change at Week 52 (n=114) | -0.1 (0.4)

15. Secondary Outcome: Change From Baseline in Insulin Level at Week 4, 12, 28 and 52
Time Frame: Baseline, Week 4, 12, 28, 52
Population: PP population. Missing values were imputed using LOCF at Week 52. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: international unit per liter (IU/L)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 107
international unit per liter (IU/L)
  Baseline (n=107) | 22.4 (27.1)
  Change at Week 4 (n=102) | -0.3 (28.9)
  Change at Week 12 (n=104) | -4.6 (20.9)
  Change at Week 28 (n=92) | -7.8 (23.5)
  Change at Week 52 (n=107) | -5.6 (31.0)

16. Secondary Outcome: Change From Baseline in the Physical Activity Index Score at Week 28 and 52
Description: Physical activity (exercise) score derived for each participant based on the frequency and intensity of physical activities: regular walking, recreational activity, cycling, and sporting activity. Six categories of total score: inactive (range: 0-2), occasional (range: 3-5), light (range: 6-8), moderate (range: 9-12), moderately vigorous (range: 13-20), and vigorous (>=21). Higher total score = higher frequency and intensity of physical activity.
Time Frame: Baseline, Week 28, 52
Population: PP population. Missing values at Week 52 were imputed using LOCF. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 112
units on a scale
  Baseline | 7.3 (6.8)
  Change at Week 28 | 0.6 (6.5)
  Change at Week 52 | 0.5 (6.3)

17. Secondary Outcome: Change From Baseline in QT Interval Corrected for Heart Rate (QTc) at Week 4, 12, 28 and 52
Description: QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. QTc is the QT interval corrected for heart rate. Corrected QT interval using Fridericia's heart rate correction formula: QTcF = QT/RR^1/3, where RR=RR interval in seconds (60 divided by heart rate).
Time Frame: Baseline, Week 4, 12, 28, 52
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study medication, had baseline and at least 1 post-baseline MS measure. Missing values at Week 52 were imputed using LOCF. N (number of participants analyzed)=participants evaluable for this measure. n=evaluable participants at specified time points.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ziprasidone
Number analyzed (Participants) | 56
milliseconds
  Baseline (n=56) | 413.2 (24.1)
  Change at Week 4 (n=4) | 0.9 (22.0)
  Change at Week 12 (n=14) | 3.4 (27.7)
  Change at Week 28 (n=38) | 6.6 (23.7)
  Change at Week 52 (n=56) | 7.6 (22.8)

18. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score, Positive and Negative Subscale Scores at Week 12, 28 and 52
Description: Assesses positive and negative symptoms, general psychopathology specifically associated with schizophrenia. Scale consists of 30 items, each rated on scale from 1 (symptom not present) - 7 (symptoms extremely severe). Sum of 30 items is defined as PANSS total score, range:30-210. 7 items make up positive scale (delusions, conceptual disorganization, hallucinatory behavior); total range: 7-49. 7 items make up negative scale (blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal); total range: 7-49. For each subscale, total score: higher score=greater severity.
Time Frame: Baseline, Week 12, 28, 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 113
units on a scale
  Baseline: Total Score (n=112) | 64.1 (17.8)
  Baseline: Positive Subscale Score (n=113) | 13.6 (4.6)
  Baseline: Negative Subscale Score (n=112) | 17.9 (6.6)
  Change at Week 12: Total Score (n=110) | -5.7 (11.6)
  Change at Week 12: Positive Subscale Score (n=112) | -1.0 (3.2)
  Change at Week 12: Negative Subscale Score (n=111) | -1.9 (4.5)
  Change at Week 28: Total Score (n=98) | -4.4 (14.3)
  Change at Week 28: Positive Subscale Score (n=100) | -0.9 (4.5)
  Change at Week 28: Negative Subscale Score (n=98) | -1.6 (5.3)
  Change at Week 52: Total Score (n=112) | -3.2 (17.0)
  Change at Week 52: Positive Subscale Score (n=113) | -0.2 (5.6)
  Change at Week 52: Negative Subscale Score (n=112) | -1.7 (5.5)

19. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Scale (CGI-S) Score at Week 12, 28 and 52
Description: CGI-S is a single-item, clinician-rated scale that assesses the global severity of the participants overall illness. CGI-S ratings range from 1 (normal, not at all ill) to 7 (among the most severely ill participants).
Time Frame: Baseline, Week 12, 28, 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 113
units on a scale
  Baseline (n=113) | 3.3 (0.9)
  Change at Week 12 (n=112) | -0.3 (0.7)
  Change at Week 28 (n=100) | -0.2 (0.8)
  Change at Week 52 (n=113) | -0.2 (1.1)

20. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Scale Score
Description: CGI-I is a single-item, clinician-rated scale that assesses global improvement in the participants clinical state in response to study treatment, and as compared to their status at pre-treatment baseline. Possible CGI-I scores range from 1 to 7, where 1=very much improved, 4=no change and 7=very much worse.
Time Frame: Endpoint (premature discontinuation or Week 52)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 107
units on a scale | 3.2 (1.4)

21. Secondary Outcome: Change From Baseline in Drug-Attitude Inventory-30-Item Scale (DAI-30) Score at Week 28 and 52
Description: DAI, a 30-item scale measuring subjective responses to medication (including acceptability and tolerability which aims to understand the factors influencing treatment adherence). Scale has 15 items (statements) scored as true and 15 items scored as false. An overall calculated score ranged from -15 to 15, where a positive score indicated a positive subjective response (compliant), a negative score indicated non-compliance.
Time Frame: Baseline, Week 28, 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 105
units on a scale
  Baseline (n=105) | -1.3 (5.8)
  Change at Week 28 (n=104) | 0.4 (6.5)
  Change at Week 52 (n=105) | -0.1 (6.1)

22. Secondary Outcome: Change From Baseline in Social and Occupational Functioning Assessment Scale (SOFAS) Score at Week 28 and 52
Description: SOFAS: a 0-100 single score scale focusing exclusively on participant's level of social and occupational functioning; not directly influenced by overall severity of participant's psychological symptoms; higher score = higher level of functioning.
Time Frame: Baseline, Week 28, 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 111
units on a scale
  Baseline | 57.2 (11.5)
  Change at Week 28 | 1.6 (11.3)
  Change at Week 52 | 1.1 (11.4)

23. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) - 5 Dimensions Index (EQ-I) Score at Week 28 and 52
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 28, 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 111
units on a scale
  Baseline | 0.8 (0.3)
  Change at Week 28 | 0.0 (0.2)
  Change at Week 52 | 0.0 (0.2)

24. Secondary Outcome: Changes From Baseline in European Quality of Life (EuroQoL) - 5 Dimensions Visual Analog Scale (VAS) Score at Week 28 and 52
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 28, 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 112
units on a scale
  Baseline (n=112) | 58.8 (27.4)
  Change at Week 28 (n=111) | 4.7 (30.5)
  Change at Week 52 (n=112) | 5.7 (30.4)

25. Secondary Outcome: Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score at Week 1, 2, 4, 8, 12, 20, 28, 36, 44 and 52
Description: C-SSRS assessed whether participant experienced following: completed suicide(1), suicide attempt(2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior(3)("Yes" on "preparatory acts or behavior"), suicidal ideation(4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act/some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior(7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline, Week 1, 2, 4, 8, 12, 20, 28, 36, 44 and 52
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 20/172
Other Adverse Events (participants affected / at risk) | 122/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=172)
Appendicitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Attention-seeking behaviour (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucinations, mixed (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 3
Schizophrenia (Psychiatric disorders) | 5
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=172)
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 21
Nasopharyngitis (Infections and infestations) | 13
Akathisia (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 15
Headache (Nervous system disorders) | 22
Somnolence (Nervous system disorders) | 17
Anxiety (Psychiatric disorders) | 33
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 50
Restlessness (Psychiatric disorders) | 10

LIMITATIONS AND CAVEATS:
The study was prematurely terminated by sponsor due to changes in organizational strategy and resources, not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.